CLINICAL TRIAL: NCT06403046
Title: Does Successive Intra-articular Injections of Tenoxicam or Meloxicam Affect Treatment Outcomes of Temporomandibular Joint Anterior Disc Displacement With Reduction? (A Randomized Controlled Trial)
Brief Title: Does Successive Intra-articular Injections of Tenoxicam or Meloxicam Affect Treatment of TMJ Displacement
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Nagi Alghandour, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 9
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Joint Disc Displacement, With Reduction
MeSH Terms: interventions — Injections, Intra-Articular; Arthrocentesis

STUDY DESIGN:
Intervention Model Description: two groups each groups consists of 15 participants & the total number of participants is 30 as the patients are divided into (Tx group) and (Mx group) after labeling them in sequential numbers
Who Masked: Care Provider, Investigator
Masking Description: An independent staff member will randomly allocate the patients into (Tx group) and (Mx group) after labeling them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Study group (Experimental): The study represents a randomized clinical trial that compares the short- and long-term effects of three repeated intraarticular injections of Tenoxicam post-arthrocentesis immediately, after one month, and two months after, with a one-month interval between each injection, for the alleviation of constitutional symptoms in patients with TMJ anterior disc displacement with reduction.
  Interventions: Drug: intraarticular injection
- The Control group (Experimental): The study represents a randomized clinical trial that compares the short- and long-term effects of three repeated intraarticular injections of Meloxicam post-arthrocentesis immediately, after one month, and two months after, with a one-month interval between each injection, for the alleviation of constitutional symptoms in patients with TMJ anterior disc displacement with reduction.
  Interventions: Drug: intraarticular injection

INTERVENTIONS:
Drug: intraarticular injection — all patients will be subjected to routine (TMJ) arthrocentesis followed by Tenoxicam injection into the superior joint space in the (Tx group) and Meloxicam injection among the patients of (Mx group).
  Other Names: arthrocentesis

SUMMARY:
The temporomandibular joint's (TMJ) articular disc, situated between the mandibular condyle's convexity and the articular tubercle's slope, is the most intricate synovial articulation in the human body. While the usual discal position as defined by magnetic resonance imaging (MRI) places the posterior discal band at the 12 o'clock position atop the mandibular condyle's maximum convexity, this discal disposition is altered in over 30% of the population without any accompanying physical symptoms. This denotes that rather than correcting the anatomical disc position, the treatment for discal displacement would primarily focus on symptom relief.

DETAILED DESCRIPTION:
Up until 1975, the only treatment options for (TMJ) internal derangement were surgical procedures that involved either repositioning the articular disc or removing it. Arthroscopic lavage was first described by Ohnishi as a way to dissolve adhesions and remove the inflammatory mediators, which reduced the pain, increased the mouth opening, and increased the harmony between the mandibular condyle and the articular disc, even though their native anatomical relation was not restored. Nitzan et al. in 1991 described arthrocentesis as a conservative method for (TMJ) lavage that discarded the arthroscopic morbidity and the need for costly tools and primarily aimed to utilize the hydraulic pressure of the lavage solution to wash out the inflammatory mediators, and release the articular disc adhesions.

The direct injection of a therapeutic agent into a joint cavity is known as intra-articular injection. Which usually aims to relieve arthralgia, suppress inflammation, and enhance joint function.

Various therapeutic agents are being deposited intra-articularly, including corticosteroids, hyaluronic acid, platelet-rich plasma and fibrin, opioids, corticosteroids, anxiolytics, muscle relaxants, antidepressants, anticonvulsants, and nonsteroidal anti-inflammatory drugs (NSAIDs).

(NSAIDs) the direct inhibition of the cyclooxygenase (COX) conversion of arachidonic acid to prostaglandins has been used to treat inflammatory articular diseases.

Oxicam-derived Tenoxicam and Meloxicam are inexpensive and readily available (NSAIDs); frequently injected intraarticularly following knee arthroscopy and (TMJ) arthrocentesis by virtue of their sustained drug delivery and long-lasting inflammatory effect.

Tenoxicam is a nonselective (NSAID) that inhibits both COX-1 and COX-2. On the other hand, Meloxicam is a selective COX-2 inhibitor.

The study aims to design a randomized controlled trial that compares the effect of intra-articular injection of the non-selective (NSAID) Tenoxicam versus the selective COX-2 inhibitor Meloxicam after arthrocentesis on alleviating the clinical signs and symptoms of (TMJ) disc displacement with reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with an age range of 18-45 years.
2. Those patients with the radiographic interpretation of unilateral or bilateral (TMJ) anterior disc displacement with reduction with the clinical signs of pain, limitation of mouth opening, and TMJ clicking; Wilkes classification type II.

Exclusion Criteria:

1. Clinical or radiographic signs of disc displacement without reduction, osteoarthritis, or articular bony changes.
2. Previous (TMJ) surgery, arthrocentesis, or occlusal splints.
3. Any systemic disease affecting the temporomandibular joint's anatomy, mechanical function, or outcome of the proposed treatment.
4. Those Patients with a history of allergic reactions to any components of the injectable solutions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Clicking | 9 months
  Absence or presence of clicking
Visual analogue scale | 9 months
  Scale from 1 to 10 which the 10 is the worst pain
Maximal interincisal opening | 9 months
  Increase in interincisal opening

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No